CLINICAL TRIAL: NCT05748119
Title: A Phase I, Double-Blind, Placebo-Controlled, Single and Multiple Oral Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MEB-1170 in Healthy Subjects
Brief Title: A Study to Assess the Safety of MEB-1170 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mebias Discovery, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MEB-1170-101
Record Dates: First submitted 2022-10-31; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (32):
- A1a Placebo (Placebo Comparator): Single Sentinel Placebo Comparator for 20 mg Dose of MEB-1170
  Interventions: Drug: Placebo
- A1a MEB-1170 (Experimental): Single MEB-1170 Sentinel 20 mg Dose
  Interventions: Drug: MEB-1170
- A1b Placebo (Placebo Comparator): Single Placebo comparator for 20 mg dose cohort of MEB-1170
  Interventions: Drug: Placebo
- A1b MEB-1170 (Experimental): Single MEB-1170 20 mg dose cohort
  Interventions: Drug: MEB-1170
- A2a Placebo (Placebo Comparator): Single Sentinel Placebo Comparator for 60 mg Dose of MEB-1170
  Interventions: Drug: Placebo
- A2a MEB-1170 (Experimental): Single MEB-1170 Sentinel 60 mg Dose
  Interventions: Drug: MEB-1170
- A2b Placebo (Placebo Comparator): Single Placebo comparator for 60 mg dose cohort of MEB-1170
  Interventions: Drug: Placebo
- A2b MEB-1170 (Experimental): Single MEB-1170 60 mg dose cohort
  Interventions: Drug: MEB-1170
- A3a Placebo (Placebo Comparator): Single Sentinel Placebo Comparator for 120 mg Dose of MEB-1170
  Interventions: Drug: Placebo
- A3a MEB-1170 (Experimental): Single MEB-1170 Sentinel 120 mg Dose
  Interventions: Drug: MEB-1170
- A3b Placebo (Placebo Comparator): Single Placebo comparator for 120 mg dose cohort of MEB-1170
  Interventions: Drug: Placebo
- A3b MEB-1170 (Experimental): Single MEB-1170 120 mg dose cohort
  Interventions: Drug: MEB-1170
- A4a Placebo (Placebo Comparator): Single Sentinel Placebo Comparator for 200 mg Dose of MEB-1170
  Interventions: Drug: Placebo
- A4a MEB-1170 (Experimental): Single MEB-1170 Sentinel 200 mg Dose
  Interventions: Drug: MEB-1170
- A4b Placebo (Placebo Comparator): Single Placebo comparator for 200 mg dose cohort of MEB-1170
  Interventions: Drug: Placebo
- A4b MEB-1170 (Placebo Comparator): Single MEB-1170 200 mg dose cohort
  Interventions: Drug: MEB-1170
- A5a Placebo (Placebo Comparator): Single Sentinel Placebo Comparator for 400 mg Dose of MEB-1170
  Interventions: Drug: Placebo
- A5a MEB-1170 (Experimental): Single MEB-1170 Sentinel 400 mg Dose
  Interventions: Drug: MEB-1170
- A5b Placebo (Placebo Comparator): Single Placebo comparator for 400 mg dose cohort of MEB-1170
  Interventions: Drug: Placebo
- A5b MEB-1170 (Experimental): Single MEB-1170 400 mg dose cohort
  Interventions: Drug: MEB-1170
- B1 Placebo (Placebo Comparator): MAD Placebo 60 mg comparator cohort of MEB-1170
  Interventions: Drug: Placebo
- B1 MEB-1170 (Experimental): MAD 60 mg MEB-1170 cohort
  Interventions: Drug: MEB-1170
- B2 Placebo (Placebo Comparator): MAD Placebo 100 mg comparator cohort of MEB-1170
  Interventions: Drug: Placebo
- B2 MEB-1170 (Experimental): MAD 100 mg MEB-1170 cohort
  Interventions: Drug: MEB-1170
- B3 Placebo (Placebo Comparator): MAD Placebo 200 mg comparator cohort of MEB-1170
  Interventions: Drug: Placebo
- B3 MEB-1170 (Experimental): MAD 200 mg MEB-1170 cohort
  Interventions: Drug: MEB-1170
- B4 Placebo (Placebo Comparator): MAD Placebo 400 mg comparator cohort of MEB-1170
  Interventions: Drug: Placebo
- B4 MEB-1170 (Experimental): MAD 400 mg MEB-1170 cohort
  Interventions: Drug: MEB-1170
- A3a Placebo Fed State (Placebo Comparator): Single Sentinel Placebo Comparator for 120 mg Dose of MEB-1170 in Fed State
  Interventions: Drug: Placebo
- A3a MEB-1170 Fed State (Experimental): Single Sentinel 120 mg Dose of MEB-1170 in Fed State
  Interventions: Drug: MEB-1170
- A3b Placebo Fed State (Placebo Comparator): Single Placebo comparator for 120 mg dose cohort of MEB-1170 in Fed State
  Interventions: Drug: Placebo
- A3b MEB-1170 Fed State (Experimental): Single MEB-1170 120 mg dose cohort in Fed State
  Interventions: Drug: MEB-1170

INTERVENTIONS:
Drug: MEB-1170 — Depending on the dosage, either 20 mg, 40 mg capsules, or a combination of both
  Arms: A1a MEB-1170; A1b MEB-1170; A2a MEB-1170; A2b MEB-1170; A3a MEB-1170; A3a MEB-1170 Fed State; A3b MEB-1170; A3b MEB-1170 Fed State; A4a MEB-1170; A4b MEB-1170; A5a MEB-1170; A5b MEB-1170; B1 MEB-1170; B2 MEB-1170; B3 MEB-1170; B4 MEB-1170
Drug: Placebo — Equivalent number and size of capsules containing placebo
  Arms: A1a Placebo; A1b Placebo; A2a Placebo; A2b Placebo; A3a Placebo; A3a Placebo Fed State; A3b Placebo; A3b Placebo Fed State; A4a Placebo; A4b Placebo; A5a Placebo; A5b Placebo; B1 Placebo; B2 Placebo; B3 Placebo; B4 Placebo

SUMMARY:
Primary Objective: To determine the safety and tolerability of single and multiple ascending oral doses of MEB-1170 in healthy subjects.

Secondary Objectives:

1. To determine the single and multiple oral dose pharmacokinetic profiles of MEB-1170 and the primary metabolite, M373, in healthy subjects.
2. To determine the effect of food on the pharmacokinetic (PK) profile of a single oral dose of MEB-1170 in healthy subjects.
3. To assess the pharmacodynamic (PD) response following single and multiple oral doses of MEB-1170

DETAILED DESCRIPTION:
Study Design: This will be a double-blind, placebo-controlled, single and multiple oral dose study conducted in two parts:

Part A: SAD+FE:

Part A will comprise a single ascending dose (SAD), sequential cohort study, incorporating a food effect (FE) evaluation. Up to 40 subjects will be studied in 5 cohorts (Cohorts A1 to A5), each cohort consisting of 8 subjects (6 treated with MEB-1170, 2 treated with placebo).

Subjects in Cohorts A1, A2, A4 and A5 will participate in 1 treatment period only, residing at the CRU from Day -1 (the day before dosing) to Day 3 (48 hours postdose). Subjects in Cohort A3 will participate in 2 treatment periods (once in fasted state, once in fed state) separated by a minimum of 6 days. All subjects will return for a poststudy visit approximately 5 to 7 days after their final dose.

Each Cohort will include sentinel dosing such that two subjects (one active and one placebo) will be dosed at least 48 hours before the remaining subjects in the cohort. Continuation to dose the remaining subjects will be at the Investigator's discretion, in consultation with the Sponsor.

All doses will be administered in accordance with a randomization schedule in the fasted state in the morning of Day 1, except for Cohort A3 Treatment Period 2 where MEB-1170 will be given 30 minutes after start of a high fat breakfast (see below). Each subject in Cohorts A1, A2, A4 and A5 will receive only a single dose of MEB-1170 or placebo during the study.

Subjects in Cohort A3 will participate in a 2-period treatment design in which they will be assessed for both the single-dose of MEB-1170 in a Fed and in a Fasted condition. Subjects will receive the same treatment (ie, either MEB-1170 or placebo) in both Period 1 and Period 2, and thus subjects will receive either two single doses of MEB-1170 or two single doses of placebo during the study. Fasting state assessments will occur in Period 1 and Fed state assessments in Period 2.

SAD Assessments:

* Safety/tolerability throughout study
* Physical examination, vital signs, clinical laboratory findings, and ECG
* PK concentrations
* PD assessments (pupillometry, capnography, oximetry, cold pressor testing)

Following the completion of each cohort, a safety and tolerability review will be conducted by the Safety Review Committee (SRC; see below) prior to proceeding to the next cohort. Based on this review, a decision may be made to continue the study as planned, repeat the same dose in another Cohort, assess a lower dose, add an intermediate dose, or terminate the study. Additionally, if no dose limiting toxicities are seen, further cohorts at higher doses may be added.

Part B: MAD:

Part B will comprise a multiple ascending dose (MAD), sequential cohort study. This part will be initiated after the first three SAD cohorts have been fully evaluated for safety and tolerability and the SRC has concluded that the MAD portion may commence. Up to 32 subjects will be studied in 4 cohorts (Cohorts B1 to B4), each cohort consisting of 8 subjects.

In each of Cohorts B1 to B4, 6 subjects will receive MEB-1170 and 2 will receive placebo. Once-daily dosing will occur on Days 1 to 7, inclusive, for all subjects. Each subject will participate in 1 treatment period only, residing at the CRU from the evening of Day -1 (the day before dosing) until the morning of Day 9 (48 hours after the final dose on Day 7).

All subjects will return for a poststudy visit 6 to 8 days after their final dose for a final safety assessment.

Dose levels to be studied will be determined following review of data from Part A. Following completion of each cohort in Part B, a safety and tolerability review will be conducted by the SRC prior to proceeding to the next cohort (see below). Based on this review, a decision may be made to continue the study as planned, repeat the same dose in another Cohort, assess a lower dose, add an intermediate dose or terminate the study. Additionally, if no dose limiting toxicities are seen, further cohorts at higher doses may be added.

MAD Assessments:

* Safety/tolerability throughout study
* Physical examinations, vital signs, clinical laboratory findings, and ECG
* PK concentration (see Schedule of Assessments for details)
* PD assessments (pupillometry, capnography, cold pressor testing, oximetry)

Reference Therapy, Dose and Mode of Administration:

Matching placebo capsule administered orally.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, subjects must meet all of the following inclusion criteria:

1. Provides written IRB-approved informed consent prior to any study procedures.
2. Male or female between 18 and 55 years old (inclusive) at the time of screening.
3. In good general health at screening, free from clinically significant unstable medical, surgical or psychiatric illness, at the discretion of the Investigator.
4. Subjects have a BMI between ≥ 18.0 and ≤ 32.0 kg/m2 at screening.
5. Vital signs (measured in supine position after a 5-minute rest) at screening:

   1. Systolic blood pressure ≥90 and ≤140 mmHg
   2. Diastolic blood pressure ≥50 and ≤ 90 mmHg
   3. Heart rate ≥45 and ≤100 bpm
   4. Temperature ≥35.5 °C and ≤ 37.5 °C
   5. Vital signs may be repeated once, within a minimum of 10 minutes of the completion of the last set of vital signs (while maintaining supine position until the repeated set of vital signs are collected), if it is suspected that falsely high or low levels have been obtained.
6. Adequate venous access to allow collection of multiple blood samples.
7. Negative Covid PCR test upon admission to the CRU.

   a. Subjects in Cohort A3 will need a second COVID test prior to admission the CRU for Period 2.
8. No relevant dietary restrictions and willingness to consume standard meals and snacks.
9. Willing to comply with all study procedures and requirements
10. Ability to tolerate the cold pressor test (determined at screening)
11. Women of childbearing potential (WOCBP) must be non-pregnant and non-lactating, and must use two acceptable, highly effective methods of contraception from screening until study completion, including the follow-up period (please see Section 9.4.2 for acceptable methods of contraception). Abstinence as a lifestyle choice is also acceptable. WOCBP must have a negative serum pregnancy test at Screening and negative urine pregnancy test at Day -1 and be willing to have additional pregnancy tests as required throughout the study. WOCBP must also use two acceptable, highly effective methods of contraception from screening until study completion, including the follow-up period and for 30 days after the last dose (please see Section 10.4.2 for acceptable methods of contraception). Women not of childbearing potential must be post menopausal for ≥12 months or be surgically sterile. Hysterectomy with retention of ovary function is permitted. Post-menopausal status will be confirmed through testing of FSH levels ≥ 40 IU/mL at screening for amenorrhoeic female subjects.
12. Male subjects must be surgically sterile (> 30 days since vasectomy per medical history or verbal confirmation), or, if engaged in sexual relations with a WOCBP, the subject and his partner must use two acceptable, highly effective methods of contraception from screening until study completion, including the follow-up period and 30 days after the last dose (please see Section 9.4.2 for acceptable methods of contraception). Abstinence as a lifestyle choice is also acceptable.

Exclusion Criteria:

To be eligible for this study, subjects must not meet any of the following exclusion criteria:

1. Pregnant or lactating at screening or baseline or planning to become pregnant (self or partner) at any time during the study, including the specified follow-up period.
2. History or presence of malignancy at screening or baseline, with the exception of adequately treated localised skin cancer (basal cell or squamous cell carcinoma) or carcinoma in-situ of the cervix.
3. Clinically significant infection within 28 days of the start of dosing, or infections requiring parenteral antibiotics within the 6 months prior to screening.
4. Clinically significant surgical procedure within 3 months of screening, at the discretion of the Investigator.
5. Currently suffering from clinically significant systemic allergic disease at screening or baseline or has a history of significant drug allergies including a history of anaphylactic reaction; allergic reaction due to any drug which led to significant morbidity.
6. Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within 3 months prior to study treatment administration; corticosteroids are permitted at the discretion of the Investigator), or exposure to any significantly immune suppressing drug within 30 days prior to screening or 5 half lives, whichever is longer.
7. History or presence at screening or baseline of a condition associated with significant immunosuppression.
8. Positive test for hepatitis C (HCV), hepatitis B (HBsAg), COVID, or human immunodeficiency virus (HIV) antibody at screening.
9. Symptoms of dysphagia at screening or baseline or known difficulty in swallowing capsules.
10. Any condition at screening or baseline (eg, chronic diarrhea, inflammatory bowel disease or prior surgery of the gastrointestinal tract) that would interfere with drug absorption or any disease or condition that is likely to affect drug metabolism or excretion, at the discretion of the Investigator.
11. History or presence at screening or baseline of clinically significant cardiac arrhythmia or congenital long QT syndrome.
12. QT interval corrected using Fridericia's formula (QTcF) > 450 msec for males or >470 msec for females.
13. Use of tobacco or nicotine containing products in the previous month prior to dosing or a positive urine cotinine test at Screening or Baseline.
14. Lack of willingness to abstain from the consumption of tobacco or nicotine-containing products throughout the duration of the study and until completion of the final Follow-up visit.
15. Regular alcohol consumption defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL glass of wine) or the subject is unwilling to abstain from alcohol for 48 h prior to admission and 48 h prior to Follow-up study visit.
16. Positive toxicology screening panel [urine test, including qualitative identification of barbiturates, tetrahydrocannabinol (THC), amphetamines, benzodiazepines, opiates and cocaine] or alcohol test (breath or urine) during Screening or at any time during the Study.
17. History of substance abuse or dependency or history of recreational IV drug use, over the last 5 years.
18. Use of any prescription drugs (other than permitted contraception) within 14 days prior to dosing or throughout the duration of the study, without prior approval of the Investigator and written approval of the CRO Medical Monitor.
19. Use of OTC medication including nonsteroidal anti-inflammatory drugs (NSAIDs), herbal remedies, supplements, or vitamins within 7 days prior to dosing. An exception to this is use of acetaminophen up to 4g/day to treat mild discomfort.
20. Use of any investigational drug or device within 30 days or 5 half-lives, whichever is longer, prior to screening.
21. Clinically significant blood loss, or blood or blood product donation >250 mL within 28 days of screening.
22. Subject is unwilling to refrain from strenuous exercise from 7 days prior to admission to the clinical trial unit until completion of the final onsite follow-up visit, where strenuous exercise is defined as a significant increase in the Subject's usual level of physical activity.
23. Any other reason that, in the opinion of the Investigator, might interfere with the evaluation required by the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for hematology | Through study completion, approximately 12 months
  Hematology parameters to be tested are:
  • Hemoglobin (HGB)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for hematology | Through study completion, approximately 12 months
  Hematology parameters to be tested are:
  • Hematocrit (HCT)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for hematology | Through study completion, approximately 12 months
  Hematology parameters to be tested are:
  • Erythrocytes (RBC)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for hematology | Through study completion, approximately 12 months
  Hematology parameters to be tested are:
  • Platelets (PLAT)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for hematology | Through study completion, approximately 12 months
  Hematology parameters to be tested are:
  • Leukocytes with differential (including Eosinophils (ESN), Neutrophils (NEUT), Basophils (BASO), Lymphocytes (LYM) and Reticulocytes (RETI)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested are:
  • C-reactive protein (CRP)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested are:
  • Urea (U)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Creatinine (CREAT)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Total Bilirubin (BILI) and Direct Bilirubin (BILIDIR)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Urate (URATE)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Albumin (ALB)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Alkaline Phosphatase (ALP)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Creatine phosphokinase (CPK)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Troponin 1 (TROP1)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Aspartate Aminotransferase (AST)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Alanine Aminotransferase (ALT)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Gamma- glutamyl transpeptidase (GGT)
Safety and Tolerability of Single Ascending Doses of MEB-1170 for Fasting SAD and MAD laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Glucose (GLU) (fasting labs only)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Sodium (Na)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Potassium (K)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Calcium (CA)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Chloride (CL)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Phosphate (PHOS)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for blood chemistry | Through study completion, approximately 12 months
  Biochemistry parameters to be tested - Bicarbonate (BICARB)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - pH (PH)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Specific Gravity (SPGRAV)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Creatinine (CREATININE)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Protein (PROT)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Ketones (KETONES)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Glucose (GLUC)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Total Bilirubin (BILI)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Occult Blood (OCCBLD)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Nitrite (NITRITE)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Urobilinogen (UROBIL)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 including clinical laboratory assessments for urine | Through study completion, approximately 12 months
  Macroscopic urinalysis parameters to be tested - Leukocytes (WBC)
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout QT
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout QTc
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout PR
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout RR
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout QRS
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout QTcF
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assessed by ECG | Through study completion, approximately 12 months
  A 12-lead ECG will be taken at the time points delineated in the study schedules. Additional ECG monitoring may be performed at other times if deemed necessary. Note that triplicate ECGs are required during SAD, while single ECGs are required during MAD. Readout QTcB
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 to assess adverse events | Through study completion, approximately 12 months
  Occurrence of all adverse events from first dose through end of study treatment and follow-up last visit will be monitored and treated as adverse events.
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 to assess suicidality risk | Through study completion, approximately 12 months
  Utilize C-SSRS to assess suicidality risks. Performed at screening and in both SAD and MAD
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assess vital signs | Through study completion, approximately 12 months
  Vital sign of oral body temperature will be measured at the time points specified in the study schedules with subjects resting for at least 5 minutes in a supine position. When the time of vital signs measurement coincides with a blood draw, the vital signs will be taken before the scheduled blood draw where possible while ensuring the blood draw is within the window specified in the protocol.
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assess vital signs | Through study completion, approximately 12 months
  Vital sign of blood pressure will be measured at the time points specified in the study schedules with subjects resting for at least 5 minutes in a supine position. When the time of vital signs measurement coincides with a blood draw, the vital signs will be taken before the scheduled blood draw where possible while ensuring the blood draw is within the window specified in the protocol.
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assess vital signs | Through study completion, approximately 12 months
  Vital sign of heart rate will be measured at the time points specified in the study schedules with subjects resting for at least 5 minutes in a supine position. When the time of vital signs measurement coincides with a blood draw, the vital signs will be taken before the scheduled blood draw where possible while ensuring the blood draw is within the window specified in the protocol.
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assess vital signs | Through study completion, approximately 12 months
  Vital sign of respiratory rate will be measured at the time points specified in the study schedules with subjects resting for at least 5 minutes in a supine position. When the time of vital signs measurement coincides with a blood draw, the vital signs will be taken before the scheduled blood draw where possible while ensuring the blood draw is within the window specified in the protocol.
Safety and Tolerability of Single and Multiple Ascending Doses of MEB-1170 assess subjects with a physical exam | Through study completion, approximately 12 months
  Complete physical examinations will be performed by a licensed physician, nurse practitioner or physician's assistant at the time points specified in the study schedules to ensure there are no changes compared to baseline assessment physical exams.

SECONDARY OUTCOMES:
To determine the single and multiple oral dose pharmacokinetic profiles of MEB-1170 and the primary metabolite, M373, in healthy subjects - AUC | Through study completion, approximately 12 months
  To evaluate the pharmacokinetics of single and multiple doses of MEB-1170 Pharmacokinetic parameters including, but not limited to area under the plasma concentration-time curve (AUC) from 0 to 24hours (AUC0-24)
  SAD phase,
  * Day 1 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 2, 24 hours
  * Day 3, 48 hours
  MAD phase
  * Day 1 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 2, 24 hours (immediately pre-dose)
  * Day 3, immediately pre-dose
  * Day 4, immediately pre-dose
  * Day 5, immediately pre-dose
  * Day 6, immediately pre-dose
  * Day 7, immediately pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 8: 24 hours and 36 hours post-Day 7 dose
  * Day 9: 48 hours post-Day 7 dose
To determine the single and multiple oral dose pharmacokinetic profiles of MEB-1170 and the primary metabolite, M373, in healthy subjects - Cmax | Through study completion, approximately 12 months
  To evaluate the pharmacokinetics of single and multiple doses of MEB-1170 Pharmacokinetic parameters including, but not limited to maximum plasma concentration (Cmax)
  SAD phase,
  * Day 1 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 2, 24 hours
  * Day 3, 48 hours
  MAD phase
  * Day 1 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 2, 24 hours (immediately pre-dose)
  * Day 3, immediately pre-dose
  * Day 4, immediately pre-dose
  * Day 5, immediately pre-dose
  * Day 6, immediately pre-dose
  * Day 7, immediately pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 8: 24 hours and 36 hours post-Day 7 dose
  * Day 9: 48 hours post-Day 7 dose
To determine the effect of food on the pharmacokinetic (PK) profile of a single oral dose of MEB-1170 in healthy subjects - AUC | Through study completion, approximately 12 months
  To evaluate the pharmacokinetics of single and multiple doses of MEB-1170 Pharmacokinetic parameters including, but not limited to area under the plasma concentration-time curve (AUC) from 0 to 24hours (AUC0-24)
  * Day 1 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 2, 24 hours
  * Day 3, 48 hours
To determine the effect of food on the pharmacokinetic (PK) profile of a single oral dose of MEB-1170 in healthy subjects - Cmax | Through study completion, approximately 12 months
  To evaluate the pharmacokinetics of single and multiple doses of MEB-1170 Pharmacokinetic parameters including, but not limited to maximum plasma concentration (Cmax)
  SAD phase,
  * Day 1 (pre-dose), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, and 16 hours
  * Day 2, 24 hours
  * Day 3, 48 hours
To assess the pharmacodynamic (PD) response of Pupillometry following single and multiple oral doses of MEB-1170 | Through study completion, approximately 12 months
  Pupil size and reactivity will be measured using a pupillometer device such as the NeuroOptics NPi-300 pupillometer. All pupillometer measurements will be made in the same windowless room, using standardized dim lighting.
  SAD: Check-in, immediately before dosing (t = 0) and at 3, 6, and 9 hours post-dose. MAD Day -1 and then on Days 2, 4, and 6, at hours ~t = 3, 6, and 9 post-dose.
To assess the pharmacodynamic (PD) response using capnography following single and multiple oral doses of MEB-1170 | Through study completion, approximately 12 months
  EtCO2 will be measured in millimeters of mercury (mm Hg) using noninvasive capnography.
  A Masimo/Philips EMMA® Capnograph (Americas Headquarters: Masimo Corporation, 52 Discovery, Irvine, CA 92618, USA) will be used with an airway adapter and subject mouthpiece. The EMMA Capnograph provides clear, continuous capnograph of carbon dioxide values, is simple, easy-to-use, with audible and visual alarm system for No Adapter, Clogged Adapter, No Breath (Apnea), Low Battery and adjustable High and Low EtCO2 alarm. Subjects will be instructed to breathe normally through the mouthpiece for 1 minute (according to the instructions provided with the capnograph).
  SAD: Check-in, immediately before dosing (t = 0) and at 3, 6, and 9 hours post-dose. MAD: Day -1 and then on Days 2, 4, and 6, at hours ~t = 3, 6, and 9 post-dose.
To assess the pharmacodynamic (PD) response using oximetry following single and multiple oral doses of MEB-1170 | Through study completion, approximately 12 months
  Oximetry measures oxygen saturation of circulating blood (SpO2). Measurements should be performed using the same finger during the course of the subjects' participation. For each time point indicated, a single SpO2 measure will be recorded.
  SAD: Check-in, immediately before dosing (t = 0) and at 3, 6, and 9 hours post-dose. MAD: Day -1 and then on Days 2, 4, and 6, at hours ~t = 3, 6, and 9 post-dose.
To assess the pharmacodynamic (PD) effect of analgesia using a Cold Pressor Test following single and multiple oral doses of MEB-1170 | Through study completion, approximately 12 months
  Subjects will be asked to place their left hand and forearm into an apparatus containing an ice bath, with the instruction to remove the arm from the water when they can no longer tolerate it. The upper limit for the duration of the test, which will not be communicated to the subjects, will be 5 minutes (300 seconds).
  SAD: 4.5 and 8.5 hours post-dose. MAD:Days 1, 3, and 5 at ~t = 3 hours post-dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit, Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No